CLINICAL TRIAL: NCT02517125
Title: Evaluation of the Contribution of Transoral Robotic-assisted Surgery Using Da Vinci Xi for Head and Neck Tumors
Acronym: TORS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A00173-46; 2015/2235 (Other: CSET number)
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

ARMS (1):
- Patients with head and neck cancer (Experimental)
  Interventions: Device: Transoral robotic-assisted surgery with Da Vinci Xi

INTERVENTIONS:
Device: Transoral robotic-assisted surgery with Da Vinci Xi

SUMMARY:
Head and Neck cancers are treated either with surgical resection followed by adjuvant radiotherapy, or with organ preservation strategies using definitive radiotherapy with or without concomitant chemotherapy. These treatments have long-time functional side effects and consequences on the quality of life. Transoral robotic surgery has been developing since 2006 by Weinstein and O'Malley in alternative to open surgery, to decrease the morbidity of the large surgical approach. The da Vinci device had the FDA approval and the CE mark in 2009 for transoral surgery of head and neck cancers, using previous generations of da Vinci. The last generation da Vinci Xi has received the FDA approval for laparoscopic surgery in april 2014 and the CE mark in june 2014 but has not been evaluated yet in transoral surgery. The objective of our study is therefore to study the feasibility of this transoral robotic surgery for head and neck cancers, using the da Vinci Xi.

ELIGIBILITY:
Inclusion Criteria:

1. Patient >/= 18
2. WHO Status 0-2
3. ENT cancer or solid tumor histologically proven regardless histology
4. All maps of the head and neck and any stage
5. surgically resectable according to clinical examination and preoperative investigations, confirmed in multidisciplinary meeting
6. Treatment:

   * First-line
   * Or after induction chemotherapy
   * Or local recurrence regardless of the previous treatment
   * Or second location in irradiated
7. Transoral exposition of tumor, assessed preoperatively during endoscopy during the balance of extension of the lesion
8. The patient must have accepted the possibility of surgical conversion open surgery
9. The patient must have been clearly informed of the study and have formulated his non-opposition to participate

Exclusion Criteria:

1. Metastasis (s) clinical or radiological remote, inaccessible (s) to a local curative treatment
2. post-treatment tumor progression and / or early recurrence < 3 months
3. Unresectable tumor by robotic transorally: bone infiltration, deep infiltration of soft tissues, unresectable lymphadenopathy
4. Contraindications to the suspension for transoral tumor Exposure: Dental fragility against-indication for cervical extension
5. Pathology against intercurrent-indicating cancer surgery
6. Pregnancy
7. Inability to submit to medical monitoring study for geographical, social or psychological.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Achievement rate of transoral robotic surgery | Assessed up to five years

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France